CLINICAL TRIAL: NCT02120079
Title: The Utility of in Vivo Confocal Microscopy (IVCM) to Assess Cellular Response and Efficacy of Long-term Topical Steroid Treatment in Patients With Dry Eye Disease (DED)
Brief Title: The Utility of IVCM to Assess Cellular Response and Efficacy of Long-term Topical Steroid Treatment in Patients With DED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-150H; NCT02106377 (obsolete NCT alias)
Record Dates: First submitted 2014-02-12; First posted 2014-04-22 (Estimated); Results first posted 2022-03-23 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Dry Eye Disease
Keywords: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Loteprednol Etabonate; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lotemax (Active Comparator): Lotemax (loteprednol etabonate) 0.5% is a prescription-only, preserved ophthalmic suspension supplied by Bausch & Lomb, Inc. Lotemax (loteprednol etabonate) 0.5% has been approved by the FDA for treatment of ocular inflammation with a maximum dosing frequency of 24 drops per eye per day. It is a C-20 ester-based corticosteroid, with a potent anti-inflammatory efficacy, but decreased impact on intraocular pressure (IOP) compared to other corticosteroids, which may increase IOP. The medication will be applied topically to both eyes for 6 weeks with the following regimen: four times a day for 2 weeks, twice daily for 2 weeks, and once daily for 2 weeks.
  Interventions: Drug: Lotemax; Diagnostic Test: In Vivo Confocal Microscopy (IVCM)
- Soothe Tired Eyes Lubricant Eye Drop (Artificial Tears) (Active Comparator): Soothe Tired Eyes Lubricant Eye Drop (Bausch & Lomb Inc.) is a preserved artificial tear which is used to relieve the dryness of the eye and to prevent further irritation. Its active ingredient is glycerin 1%. The artificial tear will be applied topically to both eyes for 6 weeks with the following regimen: four times a day for 2 weeks, twice daily for 2 weeks, and once daily for 2 weeks.
  Interventions: Drug: Soothe Tired Eyes Lubricant Eye Drop (Artificial Tears); Diagnostic Test: In Vivo Confocal Microscopy (IVCM)

INTERVENTIONS:
Drug: Lotemax — Lotemax (loteprednol etabonate) 0.5% will be applied topically to both eyes for 6 weeks with the following regimen: four times a day for 2 weeks, twice daily for 2 weeks, and once daily for 2 weeks.
  Other Names: Lotemax (loteprednol etabonate) 0.5%
  Arms: Lotemax
Drug: Soothe Tired Eyes Lubricant Eye Drop (Artificial Tears) — Soothe Tired Eyes Lubricant Eye Drop will be applied topically to both eyes for 6 weeks with the following regimen: four times a day for 2 weeks, twice daily for 2 weeks, and once daily for 2 weeks.
  Other Names: Soothe Tired Eyes Lubricant Eye Drop (Bausch & Lomb Inc.)
  Arms: Soothe Tired Eyes Lubricant Eye Drop (Artificial Tears)
Diagnostic Test: In Vivo Confocal Microscopy (IVCM) — In vivo confocal microscopy (IVCM) is a new imaging method, which allows visualization of the corneal structures at the cellular level. With a magnification of 800 times, it makes it possible to detect and quantify changes in the epithelial layers and sub-basal nerve plexus.

SUMMARY:
This research study is looking to see if in vivo confocal microscopy (IVCM) imaging can be used to confirm clinical findings (which are noted by the doctor during an eye exam) and measure the immune response to the inflammation in the subject's cornea (the front part of the eyeball).

Additionally, this study is trying to determine the effectiveness of two eye-drops, Lotemax and artificial tears, in treating the inflammation associated with DED by measuring changes in immune cells with IVCM imaging. The subject will be treated with either Lotemax (loteprednol) or artificial tears (a lubricating eye drop with no medication). Lotemax is an FDA-approved steroid eye-drop that is often used to treat inflammation associated with DED. Artificial tears are approved by the FDA for treatment of dryness associated with DED.

Thus, this study is designed to determine the effects of the administration of a topical steroid, Lotemax, over a treatment period of 6 weeks, using novel methods of detecting efficacy. In order to achieve the aforementioned goal, subjects will be prospectively randomized to one of two treatment arms - Lotemax or artificial tear. Both groups will follow the same study schedule.

DETAILED DESCRIPTION:
IVCM is a non-invasive imaging technique that images the cornea at a cellular level with 800x magnification, using a scanning laser. The laser is used to map the cornea, and will not damage or harm the subject's eye. Studies have shown that IVCM can be used to study cells and nerves within the cornea, providing a better understanding of how the cornea reacts to irritants. IVCM has recently been used by the investigator to assess the extent of eye inflammation in cases of dry eye patients.

Current steroid therapy in dry eye disease (DED) is comprised of a 2 week duration of pulse therapy, administered twice daily (to avoid adverse effects associated with long-term steroid use). This time frame is often too short to meaningfully resolve the inflammation associated with DED. DED often occurs when there is a decrease in the eye's tear production or if there is an increase in the evaporation of the tear film (a thin layer of tears that keep the eye moist). Eye irritation and inflammation (swelling) is often associated with DED because the surface of the eye is unable to maintain a normal level of moisture.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-89 years.
* Willing and able to provide written informed consent.
* Willing and able to comply with study assessments for the full duration of the study.
* In good stable overall health.
* Corneal dendritiform cell count by confocal microscopy of >=75/mm2 (13 immune cells per image)
* Diagnosis of dry eye disease based on the followings:
* Symptoms of dry eye disease such as foreign body sensation, burning, stinging, light sensitivity for at least 6 months.
* Two or more of the following objective signs:
* Schirmer test with anesthesia <10 mm at 5 minutes [mean Schirmer between eyes.
* Tear break-up time (TBUT) of <10 seconds.
* Corneal fluorescein staining of 4 (NEI grading scheme, 0-15) in at least one eye
* Lissamine green staining of the nasal and temporal conjunctiva (NEI grading scheme, 0-18) in at least one eye

Exclusion Criteria:

* Central corneal subbasal dendritic cell count by in vivo confocal microscopy of <75/mm2 in both eyes
* Active ocular allergies
* Active allergies to steroids, aminoglycosides, or benzalkonium chloride (BAK)
* History of contact lens wear within 3 months before enrollment.
* Intraocular surgery or ocular laser surgery within 3 months before enrollment.
* History of ocular infection within 3 months before enrollment.
* History of topical (for ophthalmic use) or systemic steroid treatment (Loteprednol (other than Lotemax suspension used in our study), Difluprednate, Fluorometholone, Prednisolone, Dexamethasone, Triamcinolone, Rimexolone, Medrysone) within 1 month before enrollment. In case of topical ophthalmic steroid use, a wash-out period of 1 month is required.
* History of increased intraocular pressure after using topical steroids (steroid responsive)
* Change in systemic immunosuppression medication in the past 3 months.
* History of any change in the frequency of topical cyclosporine or oral tetracycline compounds (tetracycline, doxycycline, and minocycline) within 1 month before enrollment.
* Any condition (including language barrier) that precludes subject's ability to comply with study requirements including completion of study.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-02; Primary Completion 2017-04 (Actual); Study Completion 2018-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedram Hamrah, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Groups:
- Lotemax: Lotemax (loteprednol etabonate) 0.5% is a prescription-only, preserved ophthalmic suspension. Lotemax 0.5% is FDA approved for treatment of ocular inflammation with a maximum dosing frequency of 24 drops per eye per day. It is a C-20 ester-based corticosteroid, with a potent anti-inflammatory efficacy, but decreased impact on intraocular pressure (IOP) compared to other corticosteroids, which may increase IOP. Lotemax 0.5% will be applied topically to both eyes for 6 weeks with the following regimen: four times daily for 2 weeks, twice daily for 2 weeks, and once daily for 2 weeks.
  In Vivo Confocal Microscopy (IVCM): IVCM is a new imaging method, which allows visualization of the corneal structures at the cellular level. With a magnification of 800 times, it makes it possible to detect and quantify changes in the epithelial layers and sub-basal nerve plexus.
Period: Baseline
Arm/Group | Lotemax | Soothe Tired Eyes Lubricant Eye Drop (Artificial Tears)
Started | 17; 28 eyes | 20; 34 eyes
Completed | 17; 28 eyes | 20; 34 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes
Period: 2 Weeks
Arm/Group | Lotemax | Soothe Tired Eyes Lubricant Eye Drop (Artificial Tears)
Started | 17; 28 eyes | 20; 34 eyes
Completed | 17; 28 eyes | 20; 34 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes
Period: 6 Weeks
Arm/Group | Lotemax | Soothe Tired Eyes Lubricant Eye Drop (Artificial Tears)
Started | 17; 28 eyes | 20; 34 eyes
Completed | 17; 28 eyes | 20; 34 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Lotemax | Soothe Tired Eyes Lubricant Eye Drop (Artificial Tears) | Total
Number analyzed (Participants) | 17 | 20 | 37
Number analyzed (Eyes) | 28 | 34 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.29 (12.62) | 55.35 (15.78) | 56.24 (14.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 17 | 29
  Male | 5 | 3 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Corneal immune dendritiform cell (DC) density at Baseline [Mean (Standard Deviation); unit: cells/mm^2] | 26.83 (14.98) | 34.59 (29.15) | 30.97 (23.76)
Corneal immune dendritiform cell (DC) morphology at Baseline [Mean (Standard Deviation); unit: cells/mm2] | 90.79 (16.67) | 92.29 (23.82) | 91.59 (20.64)
Corneal fluorescein staining at Baseline [Mean (Standard Deviation); unit: Score] | 3.39 (2.50) | 4.06 (3.27) | 3.76 (2.94)
Ocular Symptoms Disease Index (OSDI) at Baseline [Mean (Standard Deviation); unit: Score] | 56.93 (29.36) | 38.46 (20.34) | 47.18 (26.35)
Lissamine Green at Baseline [Mean (Standard Deviation); unit: Score] | 3.57 (2.71) | 5.74 (4.26) | 4.76 (3.78)
Intraocular Pressure (IOP) at Baseline [Mean (Standard Deviation); unit: mmHG] | 14.50 (3.18) | 14.97 (2.46) | 14.76 (2.79)
Tear Break-Up Time (TBUT) at Baseline [Mean (Standard Deviation); unit: Seconds] | 3.99 (2.18) | 4.17 (3.30) | 4.09 (2.82)
Schirmer's at Baseline [Mean (Standard Deviation); unit: mm] — Schirmer's at Baseline (mm in 10 min)
  mm | 10.44 (8.94) | 10.57 (9.35) | 10.51 (9.09)

OUTCOME MEASURES:

1. Primary Outcome: IVCM for Density of Corneal Immune Dendritiform Cells
Description: Density (in cells/mm^2) of Corneal Immune Dendritiform Cells
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: cells/mm^2
Units Other Than Participants: eyes
Arm/Group | Lotemax | Soothe Tired Eyes Lubricant Eye Drop (Artificial Tears)
Number analyzed (Participants) | 17 | 20
Number analyzed (eyes) | 28 | 34
cells/mm^2 | 9.47 (5.13) | 28.60 (26.09)

2. Primary Outcome: IVCM for Density of Corneal Immune Dendritiform Cells
Description: Density (in cells/mm^2) of corneal immune dendritiform cells
Time Frame: 6 Weeks
Measure: Mean (Standard Deviation); unit: cells/mm^2
Units Other Than Participants: eyes
Arm/Group | Lotemax | Soothe Tired Eyes Lubricant Eye Drop (Artificial Tears)
Number analyzed (Participants) | 17 | 20
Number analyzed (eyes) | 24 | 34
cells/mm^2 | 9.80 (5.10) | 34.03 (31.92)

3. Primary Outcome: IVCM for Corneal Immune Dendritiform Cell (DC) Morphology
Description: Morphology (in cells/mm^2) of Corneal Immune Dendritiform Cells
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: cells/mm^2
Units Other Than Participants: Eyes
Arm/Group | Lotemax | Soothe Tired Eyes Lubricant Eye Drop (Artificial Tears)
Number analyzed (Participants) | 17 | 20
Number analyzed (Eyes) | 28 | 34
cells/mm^2 | 109.50 (40.56) | 97.95 (30.92)

4. Primary Outcome: IVCM for Corneal Immune Dendritiform Cell (DC) Morphology
Description: Morphology (in cells/mm^2) of Corneal Immune Dendritiform Cells
Time Frame: 6 Weeks
Measure: Mean (Standard Deviation); unit: Cells/mm^2
Units Other Than Participants: Eyes
Arm/Group | Lotemax | Soothe Tired Eyes Lubricant Eye Drop (Artificial Tears)
Number analyzed (Participants) | 17 | 20
Number analyzed (Eyes) | 24 | 34
Cells/mm^2 | 102.31 (26.25) | 89.34 (24.73)

5. Secondary Outcome: Ocular Signs: Corneal Epitheliopathy
Description: Corneal Fluorescein Staining Using the National Eye Institute (NEI) Grading Scheme Minimum score-0 Maximum score-15 Higher score means worse outcome
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: Score
Units Other Than Participants: Eyes
Arm/Group | Lotemax | Soothe Tired Eyes Lubricant Eye Drop (Artificial Tears)
Number analyzed (Participants) | 17 | 20
Number analyzed (Eyes) | 28 | 34
Score | 1.86 (2.12) | 3.18 (2.55)

6. Secondary Outcome: Ocular Signs: Corneal Epitheliopathy
Description: as for outcome 5
Time Frame: 6 Weeks
Measure: Mean (Standard Deviation); unit: Score
Units Other Than Participants: Eyes
Arm/Group | Lotemax | Soothe Tired Eyes Lubricant Eye Drop (Artificial Tears)
Number analyzed (Participants) | 17 | 20
Number analyzed (Eyes) | 26 | 34
Score | 2.00 (1.98) | 3.59 (2.75)

7. Secondary Outcome: Ocular Signs: Conjunctival Epitheliopathy
Description: Conjunctival Lissamine Green Staining Using National Eye Institute (NEI) Grading Scheme Minimum score-0 Maximum score-18 Higher score means worse outcome
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: Score
Units Other Than Participants: Eyes
Arm/Group | Lotemax | Soothe Tired Eyes Lubricant Eye Drop (Artificial Tears)
Number analyzed (Participants) | 17 | 20
Number analyzed (Eyes) | 28 | 32
Score | 3.79 (3.47) | 4.50 (4.13)

8. Secondary Outcome: Ocular Signs: Conjunctival Epitheliopathy
Description: as for outcome 7
Time Frame: 6 Weeks
Measure: Mean (Standard Deviation); unit: Score
Units Other Than Participants: Eyes
Arm/Group | Lotemax | Soothe Tired Eyes Lubricant Eye Drop (Artificial Tears)
Number analyzed (Participants) | 17 | 20
Number analyzed (Eyes) | 26 | 34
Score | 2.46 (1.86) | 3.44 (3.55)

9. Secondary Outcome: Ocular Symptoms: Ocular Surface Disease Index (OSDI) Questionnaire
Description: Total Score of the Ocular Surface Disease Index (OSDI) Questionnaire Minimum score- 0 Maximum score-100 Higher score means worse outcome
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Lotemax | Soothe Tired Eyes Lubricant Eye Drop (Artificial Tears)
Number analyzed (Participants) | 17 | 19
Score | 47.25 (27.36) | 33.16 (23.55)

10. Secondary Outcome: Ocular Symptoms: Ocular Surface Disease Index (OSDI) Questionnaire
Description: as for outcome 9
Time Frame: 6 Weeks
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Lotemax | Soothe Tired Eyes Lubricant Eye Drop (Artificial Tears)
Number analyzed (Participants) | 16 | 20
Score | 46.63 (29.15) | 36.04 (23.30)

11. Secondary Outcome: Ocular Signs: Intraocular Pressure (IOP) by Measure of Applanation Tonometry
Description: Intraocular Pressure (IOP) will be measured via Applanation and the result will have these units: mmHg
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: Eyes
Arm/Group | Lotemax | Soothe Tired Eyes Lubricant Eye Drop (Artificial Tears)
Number analyzed (Participants) | 17 | 20
Number analyzed (Eyes) | 27 | 32
mmHg | 15.52 (2.87) | 14.50 (3.32)

12. Secondary Outcome: Ocular Signs: Intraocular Pressure (IOP) by Measure of Applanation Tonometry
Description: Intraocular Pressure (IOP) will be measured via Applanation and the result will have these units: mmHg
Time Frame: 6 Weeks
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: Eyes
Arm/Group | Lotemax | Soothe Tired Eyes Lubricant Eye Drop (Artificial Tears)
Number analyzed (Participants) | 17 | 20
Number analyzed (Eyes) | 26 | 34
mmHg | 16.88 (2.30) | 13.76 (3.32)

13. Secondary Outcome: Ocular Signs: Tear Break Up Time (TBUT)
Description: Tear Break Up Time (TBUT) will be recorded in seconds
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: Seconds
Units Other Than Participants: Eyes
Arm/Group | Lotemax | Soothe Tired Eyes Lubricant Eye Drop (Artificial Tears)
Number analyzed (Participants) | 17 | 20
Number analyzed (Eyes) | 28 | 32
Seconds | 5.20 (3.48) | 3.93 (1.91)

14. Secondary Outcome: Ocular Signs: Tear Break Up Time (TBUT)
Description: Tear Break Up Time (TBUT) will be recorded in seconds
Time Frame: 6 Weeks
Measure: Mean (Standard Deviation); unit: Seconds
Units Other Than Participants: Eyes
Arm/Group | Lotemax | Soothe Tired Eyes Lubricant Eye Drop (Artificial Tears)
Number analyzed (Participants) | 17 | 20
Number analyzed (Eyes) | 26 | 34
Seconds | 4.83 (3.68) | 3.44 (2.04)

15. Secondary Outcome: Ocular Signs: Schirmer's Test With Anesthesia
Description: The Schirmer's Test (performed using Anesthesia) will be measured in mm.
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Eyes
Arm/Group | Lotemax | Soothe Tired Eyes Lubricant Eye Drop (Artificial Tears)
Number analyzed (Participants) | 17 | 20
Number analyzed (Eyes) | 28 | 32
mm | 7.98 (4.98) | 6.88 (5.92)

16. Secondary Outcome: Ocular Signs: Schirmer's Test With Anesthesia
Description: The Schirmer's Test (performed using Anesthesia) will be measured in mm.
Time Frame: 6 Weeks
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Eyes
Arm/Group | Lotemax | Soothe Tired Eyes Lubricant Eye Drop (Artificial Tears)
Number analyzed (Participants) | 17 | 20
Number analyzed (Eyes) | 25 | 34
mm | 8.16 (4.78) | 8.18 (6.06)

ADVERSE EVENTS:
Time Frame: 6 Weeks
Groups:
- Lotemax: Lotemax (loteprednol etabonate) 0.5% is a prescription-only, preserved ophthalmic suspension. Lotemax (loteprednol etabonate) 0.5% has been approved by the FDA for treatment of ocular inflammation with a maximum dosing frequency of 24 drops per eye per day. It is a C-20 ester-based corticosteroid, with a potent anti-inflammatory efficacy, but decreased impact on intraocular pressure (IOP) compared to other corticosteroids, which may increase IOP. The medication will be applied topically to both eyes for 6 weeks with the following regimen: four times daily for 2 weeks, twice daily for 2 weeks, and once daily for 2 weeks.
  Lotemax: Lotemax (loteprednol etabonate) 0.5% will be applied topically to both eyes for 6 weeks with the following regimen: four times a day for 2 weeks, twice daily for 2 weeks, and once daily for 2 weeks.
  In Vivo Confocal Microscopy (IVCM): In vivo confocal microscopy (IVCM) is a new imaging method, which allows visualization of
Arm/Group | Lotemax | Soothe Tired Eyes Lubricant Eye Drop (Artificial Tears)
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/20
Other Adverse Events (participants affected / at risk) | 0/17 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT02120079/Prot_SAP_000.pdf